CLINICAL TRIAL: NCT06967454
Title: Manipulation of Whey Permeate Formulation for Better Fluid Retention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Collaborators: University of Surrey (Other)
Responsible Party: Principal Investigator, Catrin Roberts, Principle investigator, Northumbria University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: NorthumbriaU (CR/PR/2)
Record Dates: First submitted 2025-05-12; First posted 2025-05-13 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Beverage Hydration Index
MeSH Terms: interventions — Water; Diet, Fat-Restricted

STUDY DESIGN:
Intervention Model Description: Randomised, crossover design
Who Masked: Participant
Masking Description: Test beverages were presented to the participant in a dark bottle, and were not told which beverage they were consuming for each trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Beverage 1 (Experimental): Strawberry flavoured Water
  Interventions: Other: Water
- Beverage 2 (Experimental): Strawberry flavoured milk (Semi Skimmed)
  Interventions: Other: Semi-skimmed milk
- Beverage 3: Whey permeate (Experimental): Strawberry flavoured whey permeate
  Interventions: Other: Whey permeate
- 'Low drinkers' trial (Experimental): 150ml only of the strawberry water
  Interventions: Other: 'Low dose' water

INTERVENTIONS:
Other: Water — Participants will receive 600ml water with a strawberry flavour, in four equal aliquots across 30 minutes (150ml every 7.5minutes)
  Arms: Beverage 1
Other: Semi-skimmed milk — Participants will receive 600ml semi skimmed milk with a strawberry flavour, in four equal aliquots across 30 minutes (150ml every 7.5minutes)
  Arms: Beverage 2
Other: Whey permeate — Participants will receive 600ml whey permeate with a strawberry flavour, in four equal aliquots across 30 minutes (150ml every 7.5minutes)
  Arms: Beverage 3: Whey permeate
Other: 'Low dose' water — Participants will receive 150ml water with a strawberry flavour, across 30 minutes
  Arms: 'Low drinkers' trial

SUMMARY:
The main aim of this clinical trial is to compare the beverage hydration index of three different beverages in primary school-aged children.The Beverage Hydration Index (BHI), compares the hydration value of beverages against water. This study will explore the fluid retention capabilities of strawberry flavoured semi-skimmed milk, a new formulation of whey permeate based on a previous study, and water.

This study will also investigate:

* Identify the most effective beverage for hydration and the potential cognitive and mood benefits.
* To test if these beverages have any effect on gastric emptying
* To test if these beverages have any effect on blood glucose.
* To test the acceptability and palpability of semi-skimmed milk, whey permeate, and water in primary school-aged children.

Participants will:

* Take part in three four days (one for each beverage, and a 'low dose' trial, whereby participants will only consume 150ml of the water trial)
* Study day will take part between 9:00AM-12:30PM
* Participants will also record their food and fluid consumption the day before and consume a standardised breakfast before each trial.
* The beverage hydration index will be calculated as the mass of urine collected following control (water) consumption divided by the mass of urine collected following treatment.
* Blood and urine samples will be taken to measure hydration
* Breath samples will be taken for gastric emptying rate
* COMPASS (Computerised Mental Performance Assessment System), fNIRS (Functional Near Infrared Spectroscopy) and visual analogue scales (VAS) measures will be obtained to assess cognition/mood
* An ad libitum pasta meal will be consumed after the trial to measure appetite, along with blood glucose and further VAS to measure self reported hunger and fullness.
* A focus group will be held following completion of all three beverage trials, to gather participants opinion of each drink.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 9-11
* Healthy

Exclusion Criteria:

* Psychiatric, neurological or mental disorder.
* Children with any morbidity that might influence hydration status (i.e., renal/cardiovascular/metabolic disease), blood-borne illness, or if they were taking any medications that may impact fluid balance.
* Children that are lactose intolerant
* Children that have any food allergies

Ages: 9 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 13 (Actual)
Dates: Start 2025-05-20 (Actual); Primary Completion 2025-06-24 (Actual); Study Completion 2025-06-25 (Actual)

PRIMARY OUTCOMES:
Beverage Hydration Index | 0 minutes after beverage consumption
  Beverage Hydration index calculated as mass of urine collected following control (water) consumption divided by the mass of urine collected following treatment.
Beverage Hydration Index | 60 minutes after beverage consumption
  Beverage Hydration index calculated as mass of urine collected following control (water) consumption divided by the mass of urine collected following treatment.
Beverage Hydration Index | 120 minutes after beverage consumption
  Beverage Hydration index calculated as mass of urine collected following control (water) consumption divided by the mass of urine collected following treatment.

SECONDARY OUTCOMES:
Net Fluid Balance | 0 minutes after beverage consumption
  Net Fluid balance will be calculated subtracting total urine collected from total liquid consumed
Net Fluid Balance | 60 minutes after beverage consumption
  Net Fluid balance will be calculated subtracting total urine collected from total liquid consumed
Net Fluid Balance | 120 minutes after beverage consumption
  Net Fluid balance will be calculated subtracting total urine collected from total liquid consumed
Urine Osmolality | -30 minutes before beverage consumption
  Urine Osmolality will be measured in milliosmoles per kilogram of water.
Urine Osmolality | 0 minutes after beverage consumption
  Urine Osmolality will be measured in milliosmoles per kilogram of water.
Urine Osmolality | 60 minutes after beverage consumption
  Urine Osmolality will be measured in milliosmoles per kilogram of water.
Urine Osmolality | 120 minutes after beverage consumption
  Urine Osmolality will be measured in milliosmoles per kilogram of water.
Serum Osmolality | -30 minutes (before beverage consumption)
  Serum Osmolality will be measured in milliosmoles per kilogram of water.
Serum Osmolality | 0 minutes after beverage consumption
  Serum Osmolality will be measured in milliosmoles per kilogram of water.
Serum Osmolality | 30 minutes after beverage consumption
  Serum Osmolality will be measured in milliosmoles per kilogram of water.
Serum Osmolality | 60 minutes after beverage consumption
  Serum Osmolality will be measured in milliosmoles per kilogram of water.
Serum Osmolality | 120 minutes after beverage consumption
  Serum Osmolality will be measured in milliosmoles per kilogram of water.
Gastric emptying rate | -30 minutes (before beverage), 15, 30, 45, 60, 75, 90, 105, 120 minutes (after beverage consumption)
  Test beverages will be infused with 13C-sodium acetate and evaluated using the 13C breath test. Samples will be analysed to determine the ratio of 13CO2 to 12CO2. The change in this ratio from the baseline to post-beverage samples will be expressed as delta over baseline (DOB)
Cognitive function | -45 minutes (before beverage consumption)
  A collection of five cognitive tasks including choice reaction time, simple reaction time, Stroop, Picture recognition and Corsi blocks via Computerised Mental Performance Assessment System (COMPASS)
Cognitive function | 45 minutes (after beverage consumption)
  A collection of five cognitive tasks including choice reaction time, simple reaction time, Stroop, Picture recognition and Corsi blocks via Computerised Mental Performance Assessment System (COMPASS)
Cognitive function | 105 minutes (after beverage consumption)
  A collection of five cognitive tasks including choice reaction time, simple reaction time, Stroop, Picture recognition and Corsi blocks via Computerised Mental Performance Assessment System (COMPASS)
Neuroimaging | -45 minutes (before beverage consumption)
  Functional near-infrared spectroscopy (fNIRS) will monitor changes in the blood oxygenation and blood volume that are related to the human brain function. The headband will be worn whilst participants complete the cognitive tasks.
Neuroimaging | 45 minutes (after beverage consumption)
  Functional near-infrared spectroscopy (fNIRS) will monitor changes in the blood oxygenation and blood volume that are related to the human brain function. The headband will be worn whilst participants complete the cognitive tasks.
Neuroimaging | 105 minutes (after beverage consumption)
  Functional near-infrared spectroscopy (fNIRS) will monitor changes in the blood oxygenation and blood volume that are related to the human brain function. The headband will be worn whilst participants complete the cognitive tasks.
Subjective mood and appetite | -30 minutes (before beverage consumption), 0, 45, 105, 120 and 150minutes (after beverage consumption)
  Mood measured with visual analogue scale (VAS) on 100 mm horizontal lines. Additional VAS will be completed for thirst and appetite. Participants will simply mark a vertical line between the anchored terms, which they feel fittingly, represents how they are feeling at that time. For example, the happiness VAS will have the terms "very happy" printed on the right-hand side of the scale and "very sad" on the left-hand side. The hunger and thirst scales will have 'not hungry or thirsty' printed on the left-hand side and 'very hungry or thirsty' on the right-hand side. A low score will demonstrate that the child had put a mark at the 'not' end of the scale, a high score would show that the child had put a mark at the 'very' end of the scale.
Subjective beverage acceptability | 0 minutes (immediately after beverage consumption)
  Subjective beverage palatability and acceptability measured with visual analogue scale (VAS) on 100 mm horizontal lines. Participants will simply mark a vertical line between the anchored terms, which they feel fittingly, represents how they are feeling at that time. The participants will score terms "sour, sweet, salty, taste, hydrating, stomach bloating, drink again". The score of 0 will indicate they dislike and the score of 100 will indicate they like the beverages.
Ad libitum pasta meal | 120-150 minutes (after beverage consumption)
  Lunchtime food intake will be assessed from a standardised pasta meal offered ad libitum. Energy intake will be calculated based on the amount consumed and the nutritional information provided Nutritics. The meal will be weighed before and immediately after the participant finished eating.
Blood glucose | At -30, 0, 60, 120, 150 minutes (before after the ad-libitum lunch meal)
  Blood glucose concentrations will be measured instantly using the glucose oxidase method with an automated glucose analyser
Focus group | Following completion of all beverage trials, an average of 8 weeks
  After all participants have completed their trials, a focus group will be held to gather the children's options on the drinks.

CONTACTS AND LOCATIONS:
Overall Officials: Catrin Roberts, PhD, Principal Investigator — Northumbria University
Locations (1):
- Northumbria University, Newcastle upon Tyne, United Kingdom

IPD SHARING:
Plan to Share IPD: No